CLINICAL TRIAL: NCT06199804
Title: Determining The Effectiveness of Toy Hygiene Education For Hospitalized Mothers: Randomized Controlled Trial
Brief Title: Toy Hygiene Education For Hospitalized Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sibel Küçükoğlu (Other)
Collaborators: Health Institutes of Turkey (Other Government)
Responsible Party: Sponsor-Investigator, Sibel Küçükoğlu, Faculty of Nursing, Selcuk University
Organization: Selcuk University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SelcukUnı4235
Record Dates: First submitted 2023-12-27; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Children, Only; Educational Problems; Hospital Infection
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Intervention Model Description: In this study, stratified randomization method was used to determine the intervention and control groups. It is emphasized in the literature that the variables that affect children's compliance with hospital rules are affected by the education level of the mother and the age of the child. Therefore, to ensure homogeneity in the groups, they were stratified as the mother's education level (primary school, high school, university) and age group (1-3 and 4-6). In the study, randomizer.org was used to select 6-block A and B block combinations. Eligible participants were randomly assigned to experimental and control groups using the permuted block randomization method on a 1:1 basis.
Who Masked: Investigator
Masking Description: The population of the research consisted of mothers with children aged 1-3 and 4-6 who were treated as inpatients in the pediatric clinics of a public hospital in the central Anatolia region of Turkey between January and August 2023.
  Inclusion Criteria;
  * Mothers with children in the play (1-3) and preschool (4-6) periods
  * Those who keep toys (plastic, metal, wooden, technological) with their children
  * Mothers who are always with their children as companions
  * Mothers whose children receive inpatient treatment for at least 3 days Exclusion Criteria;
  * Mother has hearing, vision or mental problems
  * The mother has been diagnosed with OCD (Obsessive Compulsive Disorder) or has an obsession with cleaning.
  * Not being able to speak Turkish
  * Being under 18 years of age
  * Do not place the child in isolation (contact isolation, droplet isolation, respiratory isolation).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): A program was created to be given to the mothers in the experimental group in line with the content of the "Toy Hygiene Guide Book" prepared by the researchers.
  Interventions: Behavioral: Toy Hygiene Training
- Control Group (No Intervention): The researcher did not apply anything other than the clinical routine to the control group during the first three days of hospitalization.

INTERVENTIONS:
Behavioral: Toy Hygiene Training — The training was given to the mothers in 2 sessions (morning and afternoon), each lasting approximately 30 minutes, accompanied by the Toy Hygiene Guide. The sessions were presented face to face in the mother's room in the form of explaining, showing, question and answer and power point, at a time convenient for the mother and the child, outside the morning and afternoon treatment and care hours. After the first session was completed, an appointment was made with the mother for the afternoon session. In the second session, the information in the book that was not given in the first session was presented to the mothers face to face in the mother's room, outside the treatment and care hours, at a time convenient for the mother and the child. After the training was completed, a final five-minute discussion was held with the mothers in the form of a general question and answer session. The training book was given to the mothers in the experimental group on the first day.
  Arms: Experimental Group

SUMMARY:
The present study aims to evaluate the effectiveness of toy hygiene education given to mothers of hospitalized children on their knowledge and practices, as well as the cleanliness of toy surfaces.

DETAILED DESCRIPTION:
While studies show that toys contain significant amounts of pathogenic microorganisms and may be effective in the spread of hospital-acquired infections, it appears that the literature and hospital practices on the disinfection of these toys are quite limited. Additionally, there is no routine practice to ensure toy hygiene in most health institutions. Therefore, in order to prevent the transfer of infectious agents through toys, policies and guidelines regarding toy cleaning methods and frequency should be established in hospitals. At the same time, families should be educated about the fact that toys can be a source of infection, and correct behavioral changes regarding toy hygiene should be created. When the literature was examined, it was determined that there were no routine hygiene practices regarding the cleaning of toys in children's clinics in Turkey. For this reason, the study will examine the effect of the toy hygiene education created by the researchers on the knowledge levels and practices of mothers and the surface cleaning of toys. It is thought that the results of the study will be a basis for creating clinical guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Mothers with children in the play (1-3) and preschool (4-6) periods
* Those who keep toys (plastic, metal, wooden, technological) with their children
* Mothers who are always with their children as companions
* Mothers whose children receive inpatient treatment for at least 3 days

Exclusion Criteria:

* Mother has hearing, vision or mental problems
* The mother has been diagnosed with OCD (Obsessive Compulsive Disorder) or has an obsession with cleaning.
* Not being able to speak Turkish
* Being under 18 years of age
* Do not place the child in isolation (contact isolation, droplet isolation, respiratory isolation).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Since mothers stayed with their children, only mothers were included in the study.
Enrollment: 48 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-12-13 (Actual)

PRIMARY OUTCOMES:
Sociodemographic Questionnaire | First measurement-First day of hospitalization
  Demographic data for the mother and her sick child were questioned in the form prepared by the researchers in line with the literature (Avila-Aguero et al. 2004; Merriman et al. 2002, Deshpande et al. 2020). As variables related to the mother, age, family type, number of children, education level, employment status, perception of economic situation, place of residence and the status of receiving information about toy hygiene were questioned. For the child; It was composed of questions asking age, gender, medical diagnosis, presence of chronic disease, hospitalization, room type, and hospitalization experience.
Toy Hygiene Information Form | First measurement-First day of hospitalization
  The toy hygiene information form, prepared by the researchers in line with the literature (Avila-Aguero et al. 2004; Yokoe et al. 2009), was composed of two parts. In the first part, the types of toys that parents prefer to buy for their children, their preference for buying cleanable toys, the situation of cleaning toys before bringing them to the hospital, their practices to ensure toy hygiene in the hospital environment, and the difficulties they experience in ensuring toy hygiene in the hospital environment are questioned. In the second part of the form, a knowledge test consisting of 31 items was prepared to determine the knowledge level of mothers regarding toy hygiene. The second part of the form is answered as true or false. A high score from the knowledge test is interpreted as a high level of "toy hygiene knowledge".
Toy Surface Cleaning Level Record Form | First measurement-First day of hospitalization
  This form was created by researchers to record the level of surface cleanliness by taking a swab from the toy surface with the 3M™ Clean-Trace™ ATP device before and after the training.

SECONDARY OUTCOMES:
Toy Hygiene Information Form | Second measurement-Third day of hospitalization
  The toy hygiene information form, prepared by the researchers in line with the literature (Avila-Aguero et al. 2004; Yokoe et al. 2009), was composed of two parts. In the first part, the types of toys that parents prefer to buy for their children, their preference for buying cleanable toys, the situation of cleaning toys before bringing them to the hospital, their practices to ensure toy hygiene in the hospital environment, and the difficulties they experience in ensuring toy hygiene in the hospital environment are questioned. In the second part of the form, a knowledge test consisting of 31 items was prepared to determine the knowledge level of mothers regarding toy hygiene. The second part of the form is answered as true or false. A high score from the knowledge test is interpreted as a high level of "toy hygiene knowledge".
  Only the second part of the form was remeasured.
Toy Surface Cleaning Level Record Form | Second measurement-Third day of hospitalization
  This form was created by researchers to record the level of surface cleanliness by taking a swab from the toy surface with the 3M™ Clean-Trace™ ATP device before and after the training.

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Küçükoğlu, Prof, Study Director — Selcuk University
Locations (1):
- Selcuk University, Konya, Selcuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be shared after the article is published

REFERENCES:
- [Background] Deshpande A, Dunn AN, Fox J, Cadnum JL, Mana TSC, Jencson A, Fraser TG, Donskey CJ, Gordon SM. Monitoring the effectiveness of daily cleaning practices in an intensive care unit (ICU) setting using an adenosine triphosphate (ATP) bioluminescence assay. Am J Infect Control. 2020 Jul;48(7):757-760. doi: 10.1016/j.ajic.2019.11.031. Epub 2019 Dec 26. PMID 31883729
- [Background] Yokoe D, Casper C, Dubberke E, Lee G, Munoz P, Palmore T, Sepkowitz K, Young JA, Donnelly JP; Center for International Blood and Marrow Transplant Research; National Marrow Donor Program; European Blood and Marrow Transplant Group; American Society of Blood and Marrow Transplantation; Canadian Blood and Marrow Transplant Group; Infectious Disease Society of America; Society for Healthcare Epidemiology of America; Association of Medical Microbiology and Infectious Diseases Canada; Centers for Disease Control and Prevention. Infection prevention and control in health-care facilities in which hematopoietic cell transplant recipients are treated. Bone Marrow Transplant. 2009 Oct;44(8):495-507. doi: 10.1038/bmt.2009.261. No abstract available. PMID 19861984
- [Result] Avila-Aguero ML, German G, Paris MM, Herrera JF; Safe Toys Study Group. Toys in a pediatric hospital: are they a bacterial source? Am J Infect Control. 2004 Aug;32(5):287-90. doi: 10.1016/j.ajic.2003.10.018. PMID 15292894
- [Result] Merriman E, Corwin P, Ikram R. Toys are a potential source of cross-infection in general practitioners' waiting rooms. Br J Gen Pract. 2002 Feb;52(475):138-40. PMID 11885823